CLINICAL TRIAL: NCT02239640
Title: Systematic Evaluation of Patients Treated With Stroke Devices for Acute Ischemic Stroke (STRATIS) Registry
Status: Completed | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-SFR005
Record Dates: First submitted 2014-09-08; First posted 2014-09-15 (Estimated); Results first posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medtronic NV market-released device: Patients experiencing an acute ischemic stroke due to a large vessel occlusion treated with a Medtronic Neurovascular market-released neurothrombectomy device.

SUMMARY:
The purpose of this registry is to assess clinical outcomes, and different factors that may affect these clinical outcomes such as systems of care, associated with the use of Covidien market-released neurothrombectomy devices intended to restore blood flow in patients experiencing acute ischemic stroke due to large intracranial vessel occlusion.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, observational registry of acute ischemic stroke patients that have or will undergo treatment with the use of a Covidien market-released neurothrombectomy device (as the initial device used to remove the thrombus) within 8 hours of stroke symptom onset, at the discretion of the investigator and independent of participation in this registry. This registry may enroll up to 1000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient or patient's legally authorized representative has given Informed Consent according to Good Clinical Practices (GCP) and/or IRB and/or local or institutional policies.
* Patient has experienced an acute ischemic stroke due to large intracranial vessel occlusion (with associated symptoms) and has been or will be treated with a Covidien market-released neurothrombectomy device, as the initial device used to remove the thrombus.
* Treatment within 8 hours of stroke onset.
* Pre-Stroke Modified Rankin Scale (mRS) score ≤ 1 (immediately) prior to stroke onset.
* Pre-treatment National Institutes of Health Stroke Scale (NIHSS) ≥ 8 and ≤ 30.

Exclusion Criteria:

* Concurrent participation in a multicenter randomized study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute Ischemic Stroke Patients
Sampling Method: Non-Probability Sample
Enrollment: 984 (Actual)
Dates: Start 2014-08-21 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nils Mueller-Kronast, M.D., Principal Investigator — Advanced Neuroscience Network/Tenet South Florida
Locations (55):
- United States (55):
  - Banner University Medical Center, Phoenix, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - University of California Irvine, Irvine, California
  - University of California Los Angeles, Los Angeles, California
  - Mercy San Juan Medical Center/ Mercy General, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Los Robles Medical Center, Thousand Oaks, California
  - Advanced Neuroscience Network/Tenet South Florida, Delray Beach, Florida
  - South Broward Hospital, Hollywood, Florida
  - Baptist Medical Center - Jacksonville, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - WellStar Kennestone Regional Medical Center, Marietta, Georgia
  - Presence St. Joseph Medical Center, Joliet, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Baptist Health Lexington/Central Baptist, Lexington, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky
  - Baptist Hospital Louisville, Louisville, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St. John Providence Hospital, Detroit, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - St. Dominic's - Jackson Memorial Hospital, Jackson, Mississippi
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Buffalo General Medical Center, Buffalo, New York
  - Crouse Hospital, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University Hospital, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Valley Baptist Medical Center, Harlingen, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Hospital, Houston, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - West Virginia University/ Ruby Memorial, Morgantown, West Virginia
  - Aurora Hospital, Milwaukee, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Only multi center data will be available

REFERENCES:
- [Derived] Jahan R, Liebeskind DS, Zaidat OO, Mueller-Kronast NH, Froehler MT, Saver JL. Stent Retriever Thrombectomy for Anterior vs. Posterior Circulation Ischemic Stroke: Analysis of the STRATIS Registry. Front Neurol. 2021 Aug 23;12:706130. doi: 10.3389/fneur.2021.706130. eCollection 2021. PMID 34504469
- [Derived] Jumaa MA, Castonguay AC, Salahuddin H, Jadhav AP, Limaye K, Farooqui M, Zaidi SF, Mueller-Kronast N, Liebeskind DS, Zaidat OO, Ortega-Gutierrez S. Middle Cerebral Artery M2 Thrombectomy in the STRATIS Registry. Stroke. 2021 Nov;52(11):3490-3496. doi: 10.1161/STROKEAHA.120.033951. Epub 2021 Jul 27. PMID 34311566
- [Derived] Zaidat OO, Liebeskind DS, Jadhav AP, Ortega-Gutierrez S, Nguyen TN, Haussen DC, Yavagal DR, Froehler MT, Jahan R, Nogueira RG, Yao TL, Alenzi BA, Bushnaq S, Mueller-Kronast NH. Impact of Age and Alberta Stroke Program Early Computed Tomography Score 0 to 5 on Mechanical Thrombectomy Outcomes: Analysis From the STRATIS Registry. Stroke. 2021 Jul;52(7):2220-2228. doi: 10.1161/STROKEAHA.120.032430. Epub 2021 Jun 3. PMID 34078106
- [Derived] Mueller-Kronast N, Froehler MT, Jahan R, Zaidat O, Liebeskind D, Saver JL; STRATIS Investigators. Impact of EMS bypass to endovascular capable hospitals: geospatial modeling analysis of the US STRATIS registry. J Neurointerv Surg. 2020 Nov;12(11):1058-1063. doi: 10.1136/neurintsurg-2019-015593. Epub 2020 May 8. PMID 32385089
- [Derived] Zaidat OO, Mueller-Kronast NH, Hassan AE, Haussen DC, Jadhav AP, Froehler MT, Jahan R, Ali Aziz-Sultan M, Klucznik RP, Saver JL, Hellinger FR Jr, Yavagal DR, Yao TL, Gupta R, Martin CO, Bozorgchami H, Kaushal R, Nogueira RG, Gandhi RH, Peterson EC, Dashti S, Given CA 2nd, Mehta BP, Deshmukh V, Starkman S, Linfante I, McPherson SH, Kvamme P, Grobelny TJ, Hussain MS, Thacker I, Vora N, Chen PR, Monteith SJ, Ecker RD, Schirmer CM, Sauvageau E, Chebl AB, Derdeyn CP, Maidan L, Badruddin A, Siddiqui AH, Dumont TM, Alhajeri A, Taqi MA, Asi K, Carpenter J, Boulos A, Jindal G, Puri AS, Chitale R, Deshaies EM, Robinson D, Kallmes DF, Baxter BW, Jumaa M, Sunenshine P, Majjhoo A, English JD, Suzuki S, Fessler RD, Delgado-Almandoz J, Martin JC, Liebeskind DS; STRATIS Investigators. Impact of Balloon Guide Catheter Use on Clinical and Angiographic Outcomes in the STRATIS Stroke Thrombectomy Registry. Stroke. 2019 Mar;50(3):697-704. doi: 10.1161/STROKEAHA.118.021126. PMID 30776994
- [Derived] Zaidat OO, Haussen DC, Hassan AE, Jadhav AP, Mehta BP, Mokin M, Mueller-Kronast NH, Froehler MT. Impact of Stent Retriever Size on Clinical and Angiographic Outcomes in the STRATIS Stroke Thrombectomy Registry. Stroke. 2019 Feb;50(2):441-447. doi: 10.1161/STROKEAHA.118.022987. PMID 30626287
- [Derived] Froehler MT, Saver JL, Zaidat OO, Jahan R, Aziz-Sultan MA, Klucznik RP, Haussen DC, Hellinger FR Jr, Yavagal DR, Yao TL, Liebeskind DS, Jadhav AP, Gupta R, Hassan AE, Martin CO, Bozorgchami H, Kaushal R, Nogueira RG, Gandhi RH, Peterson EC, Dashti SR, Given CA 2nd, Mehta BP, Deshmukh V, Starkman S, Linfante I, McPherson SH, Kvamme P, Grobelny TJ, Hussain MS, Thacker I, Vora N, Chen PR, Monteith SJ, Ecker RD, Schirmer CM, Sauvageau E, Abou-Chebl A, Derdeyn CP, Maidan L, Badruddin A, Siddiqui AH, Dumont TM, Alhajeri A, Taqi MA, Asi K, Carpenter J, Boulos A, Jindal G, Puri AS, Chitale R, Deshaies EM, Robinson DH, Kallmes DF, Baxter BW, Jumaa MA, Sunenshine P, Majjhoo A, English JD, Suzuki S, Fessler RD, Delgado Almandoz JE, Martin JC, Mueller-Kronast NH; STRATIS Investigators. Interhospital Transfer Before Thrombectomy Is Associated With Delayed Treatment and Worse Outcome in the STRATIS Registry (Systematic Evaluation of Patients Treated With Neurothrombectomy Devices for Acute Ischemic Stroke). Circulation. 2017 Dec 12;136(24):2311-2321. doi: 10.1161/CIRCULATIONAHA.117.028920. Epub 2017 Sep 24. PMID 28943516
- [Derived] Mueller-Kronast NH, Zaidat OO, Froehler MT, Jahan R, Aziz-Sultan MA, Klucznik RP, Saver JL, Hellinger FR Jr, Yavagal DR, Yao TL, Liebeskind DS, Jadhav AP, Gupta R, Hassan AE, Martin CO, Bozorgchami H, Kaushal R, Nogueira RG, Gandhi RH, Peterson EC, Dashti SR, Given CA 2nd, Mehta BP, Deshmukh V, Starkman S, Linfante I, McPherson SH, Kvamme P, Grobelny TJ, Hussain MS, Thacker I, Vora N, Chen PR, Monteith SJ, Ecker RD, Schirmer CM, Sauvageau E, Abou-Chebl A, Derdeyn CP, Maidan L, Badruddin A, Siddiqui AH, Dumont TM, Alhajeri A, Taqi MA, Asi K, Carpenter J, Boulos A, Jindal G, Puri AS, Chitale R, Deshaies EM, Robinson DH, Kallmes DF, Baxter BW, Jumaa MA, Sunenshine P, Majjhoo A, English JD, Suzuki S, Fessler RD, Delgado Almandoz JE, Martin JC, Haussen DC; STRATIS Investigators. Systematic Evaluation of Patients Treated With Neurothrombectomy Devices for Acute Ischemic Stroke: Primary Results of the STRATIS Registry. Stroke. 2017 Oct;48(10):2760-2768. doi: 10.1161/STROKEAHA.117.016456. Epub 2017 Aug 22. PMID 28830971

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Randomized: Observation registry.
Period: Overall Study
Arm/Group | Non-Randomized
Started | 984
Completed | 767
Not Completed | 217
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 72
Not completed — Death | 142

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects enrolled
Arm/Group | Overall Study
Number analyzed (Participants) | 984
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (14.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 451
  Male | 533
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Revascularization With mTICI Grades 2b-3
Description: Assess revascularization using modified Thrombolysis in Cerebral Infarction (mTICI) score at the end of the procedure. This scale determines the response of therapy for ischemic stroke based on angiographic appearances of the treated occluded vessel and the distal branches.
  Classification:
  grade 0: no perfusion grade 1: antegrade reperfusion past the initial occlusion, but limited distal branch filling with little or slow distal reperfusion grade 2a: antegrade reperfusion of less than half of the occluded target artery previously ischemic territory grade 2b: antegrade reperfusion of more than half of the previously occluded target artery ischemic territory grade 3: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches (higher values represent better outcomes)
Time Frame: Day 0-At the completion of the thrombectomy procedure
Population: 824 participants contributed to this analysis
Measure: Count of Participants; unit: Participants
Groups:
- Successful Revascularization: Successful reperfusion (mTICI 2b-3) per imaging core lab
Arm/Group | Successful Revascularization
Number analyzed (Participants) | 824
Participants | 724

2. Secondary Outcome: Incidence of Neurological Events of Interest
Description: Evaluate events causing neurological deterioration (defined as ≥ 4 worsening points from baseline on the NIHSS scale)
Time Frame: up to 90 days post index procedure
Measure: Count of Participants; unit: Participants
Groups:
- Neurological Deterioration: Neurological Deterioration up to 90 days (any event causing neurological deterioration; defined as ≥ 4 points worsening from baseline on the NIHSS scale).
Arm/Group | Neurological Deterioration
Number analyzed (Participants) | 984
Participants | 91

3. Other Pre Specified Outcome: All-cause Mortality
Time Frame: up to 90 days post index procedure
Measure: Count of Participants; unit: Participants
Groups:
- All-cause Mortality: All cause mortality up to 90 days post index stroke procedure
Arm/Group | All-cause Mortality
Number analyzed (Participants) | 984
Participants | 142

4. Other Pre Specified Outcome: Number of Participants With Good Functional Outcome (mRS 0-2)
Description: Score based on modified Rankin Scale (mRS). The modified Rankin Scale (mRS) is a scale used to measure the degree of disability or dependence in daily activities of people who has had a stroke.
  Clasiffication:
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead. (lower values represent less disability)
Time Frame: 90 days post index procedure
Population: 906 participants contributed to this analysis
Measure: Count of Participants; unit: Participants
Groups:
- mRS at 90 Days: mRS (0-2) at 90 Days
Arm/Group | mRS at 90 Days
Number analyzed (Participants) | 906
Participants | 512

5. Other Pre Specified Outcome: Incidence of Device Related Serious Adverse Events
Description: Any device-related serious adverse events associated with the use of a Covidien/Medtronic market-released neurothrombectomy device during the index stroke procedure up to 90 days post index stroke procedure.
Time Frame: up to 90 days post index procedure
Measure: Count of Participants; unit: Participants
Groups:
- Study Device-related SAEs (Site Reported): Incidence of study device-related SAEs <= 90 days post procedure
Arm/Group | Study Device-related SAEs (Site Reported)
Number analyzed (Participants) | 984
Participants | 2

6. Other Pre Specified Outcome: Time to Revascularization
Description: Arterial access puncture to revascularization measured in minutes. Lower values indicate shorter time to revascularization and vice versa.
Time Frame: Day 0-At the completion of the thrombectomy procedure
Population: 939 patients were analyzed
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Time to Revascularization: Puncture to TICI 2b-3 or completion
Arm/Group | Time to Revascularization
Number analyzed (Participants) | 939
minutes | 45.6 (29.0)

7. Other Pre Specified Outcome: Incidence of Procedure Related Serious Adverse Events
Description: Any procedure related serious adverse events occurring upon insertion of a Covidien/Medtronic market-released neurothrombectomy device during the index stroke procedure up to 90 days post index stroke procedure.
Time Frame: up to 90 days post index procedure
Measure: Count of Participants; unit: Participants
Groups:
- Procedure-related SAEs (Site Reported): Incidence of procedure-related SAEs <= 90 days post procedure
Arm/Group | Procedure-related SAEs (Site Reported)
Number analyzed (Participants) | 984
Participants | 17

ADVERSE EVENTS:
Time Frame: Up to 90 days post index stroke procedure
Description: Per protocol SAEs were collected up to 90 days post index stroke procedure: all-cause mortality, device-related SAE associated with the use of Covidien/Medtronic market-released neurothrombectomy device during the index stroke procedure and procedure related SAE occurring upon insertion of Covidien/Medtronic market-released neurothrombectomy device during the index stroke procedure. Non-SAEs were not required to be collected per protocol.
Groups:
- Adverse Events: Serious adverse events reported per protocol during the study
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 142/984
Serious Adverse Events (participants affected / at risk) | 19/984
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=984)
Cartotid Artery Dissection (Nervous system disorders) | 1 (1) — Study device-related SAE
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) — Study device-related SAE
Arteriovenous fistula (Vascular disorders) | 1 (1) — Index procedure-related SAE
Carotid artery dissection (Nervous system disorders) | 2 (2) — Index procedure-related SAE
Cerebral haemorrhage (Nervous system disorders) | 3 (3) — Index procedure-related SAE
Femoral artery dissection (Vascular disorders) | 1 (1) — Index procedure-related SAE
Headache (Nervous system disorders) | 1 (1) — Index procedure-related SAE
Hypotension (Vascular disorders) | 1 (1) — Index procedure-related SAE
Neurological decompensation (Nervous system disorders) | 1 (1) — Index procedure-related SAE
Peripheral artery thrombosis (Vascular disorders) | 1 (1) — Index procedure-related SAE
Peripheral vascular disorder (Vascular disorders) | 1 (1) — Index procedure-related SAE
Stroke in evolution (Nervous system disorders) | 3 (3) — Index procedure-related SAE
Subarachnoid haemorrhage (Nervous system disorders) | 5 (5) — Index procedure-related SAE
Unresponsive to stimuli (Nervous system disorders) | 1 (1) — Index procedure-related SAE
Vasospasm (Vascular disorders) | 1 (1) — Index procedure-related SAE
Vessel perforation (Vascular disorders) | 1 (1) — Index procedure-related SAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Researchers may Publish their individual site experience, but Sponsor reserves the exclusive right to Publish (or coordinate the Publication of) the complete accumulated results of the Registry, and to establish authorship criteria for such Publications for the Registry group based on Registry conduct and compliance, contribution to the Registry's design, management or enrollment and willingness to accept the rights and responsibilities of an author.